CLINICAL TRIAL: NCT01359670
Title: Functional Muscle Ischemia and PDE5A Inhibition in Duchenne Muscular Dystrophy
Brief Title: Tadalafil and Sildenafil for Duchenne Muscular Dystrophy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Parent Project Muscular Dystrophy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PPMD
Record Dates: First submitted 2011-05-23; First posted 2011-05-25 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2018-04

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne; muscular dystrophy; tadalafil; sildenafil; muscle ischemia; exercise
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies; Motor Activity | interventions — Tadalafil; Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tadalafil (Experimental)
  Interventions: Drug: Tadalafil
- Sildenafil (Experimental)
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Tadalafil — Escalating dose (0.25 mg/kg, 0.5 mg/kg, 1.0 mg/kg; once daily) over 2 weeks
  Other Names: Cialis; Adcirca
  Arms: Tadalafil
Drug: Sildenafil — Escalating dose (0.25 mg/kg, 0.5 mg/kg, 1.0 mg/kg; four times daily) over 2 weeks
  Other Names: Viagra; Revatio
  Arms: Sildenafil

SUMMARY:
This study, supported by Parent Project Muscular Dystrophy, will determine if tadalafil or sildenafil can improve muscle blood flow during exercise in boys with Duchenne muscular dystrophy.

DETAILED DESCRIPTION:
Duchenne muscular dystrophy (DMD) is a rare, progressive and fatal muscle disease affecting boys and accounts for 80% of muscular dystrophy cases. Tadalafil and sildenafil are medications approved by the FDA for the treatment of erectile dysfunction and pulmonary hypertension. This class of medication improves muscle blood flow in a mouse model of muscular dystrophy, but their benefit to boys with DMD is unknown. The purpose of this study is to 1) determine if tadalafil or sildenafil can improve muscle blood flow during exercise in boys with DMD; and 2) to inform the design of a subsequent, randomized, multi-center trial with clinical endpoints.

The investigators will enroll boys with DMD between the ages of 7 and 15 years who are ambulatory and without clinical heart failure. Participants will undergo 6 visits over the course of 5 weeks. The initial visit will include a medical history, physical exam, echocardiogram, and blood draw to determine eligibility for the study. Boys will be given a Holter monitor (a heart monitor) to wear for 48 hours to observe any irregular heartbeats or abnormalities.

Eligible boys will be randomized to one of the two study drugs: tadalafil or sildenafil. The boys will take a low dose (0.25mg/kg) of the study drug for the first 2 days and an intermediate dose (0.5mg/kg) for the subsequent 5 days. Then, boys will take a higher dose (1.0mg/kg) of the study drug for 1 week. Tadalafil will be taken once daily and sildenafil will be taken four times daily.

Study visits will occur 2 times at baseline, 2 times during the medication, and 1 time after washout of the medication. For these visits, boys will undergo an arm blood flow and hand grip exercise protocol. In this procedure, blood flow and oxygen delivery to the forearm muscles will be measured (noninvasively) before and during application of lower body negative pressure at rest and during handgrip exercise. Lower body negative pressure stimulates the blood flow changes that normally occur when a person sits up after lying down. During these visits, boys will complete a quality of life questionnaire, echocardiogram, and 6-minute walk tests. At home, boys will wear an accelerometer to measure physical activity and a Holter monitor to check for irregular heartbeats.

For boys who wish to continue with the study, there will be an option to cross-over and complete study visits with the drug they did not originally receive.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of DMD confirmed by muscle biopsy or DNA analysis
2. Age 7-15y
3. Ambulatory
4. No clinical evidence of heart failure

Exclusion Criteria:

1. Hypertension, diabetes, or heart failure by standard clinical criteria
2. Elevated BNP level (>100 pg/ml)
3. LVEF < 50%
4. Wheelchair bound
5. Cardiac rhythm disorder, specifically: rhythm other than sinus, SVT, atrial fibrillation, ventricular tachycardia
6. Continuous ventilatory support
7. Liver disease
8. Renal impairment
9. Contraindications to tadalafil or sildenafil (use of nitrates, alpha-blockers, CYP3A inhibitors, amlodipine, or other PDE5A inhibitors)

Ages: 7 Years to 15 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2011-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Functional muscle ischemia | For 5 study visits
  Measured by the decrease in muscle tissue oxygenation (near infrared spectroscopy) and blood flow (Doppler ultrasound) evoked by reflex sympathetic activation in exercising forearm muscle.

SECONDARY OUTCOMES:
Cardiac Function | For 5 study visits
  Echocardiogram
EKG Monitoring | 5 times over about 6 weeks
  48 hour Holter monitoring
6 Minute Walk Test | For 5 study visits
Physical Activity | 5 times over about 6-weeks
  Assessed by accelerometers
Quality of Life | For 5 study visits
  PedsQL inventory

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Victor, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States